CLINICAL TRIAL: NCT05161117
Title: Creating a Safe Inpatient Environment-Can Virtual Reality Fall Education Change Caregiver's Attitudes and Behaviors?
Brief Title: Virtual Reality Fall Education for Caregivers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The original principal investigator had an illness and then retired. After reorganization of research team, the study was changed to a single group pretest posttest design for feasibility.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Rose Hosler, Healing Solutions Coordinator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-247
Record Dates: First submitted 2021-10-08; First posted 2021-12-16 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Accidental Fall; Nurse's Role

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality education (Experimental): The experimental group will receive both an online fall prevention education module and additional education using a virtual reality simulation app for mobile devices designed for specifically for hospital caregivers
  Interventions: Behavioral: Virtual reality simulation app for caregiver education; Behavioral: online fall prevention education module
- online education only (Active Comparator): The control group will receive an online fall prevention education module
  Interventions: Behavioral: online fall prevention education module

INTERVENTIONS:
Behavioral: Virtual reality simulation app for caregiver education — Using a virtual reality headset/goggles, caregivers will engage with an interactive app experience to identify and mediate fall risk hazards in the inpatient care environment. The app will present a hospital bedroom and bathroom laden with fall risks. As the caregiver progresses through the experience, the caregiver will ambulate (virtually) through the environment with the goal of identifying fall risks inherent within that inpatient setting. Fall risks will be targeted and identified using the app "sighting" function and after focusing on the fall risk for the allotted "marking" time, will "self-resolve."
  Arms: virtual reality education
Behavioral: online fall prevention education module — Participants in both intervention and control groups will complete a 20 minute online module: Management of the Patient at Risk for Falls, through the MyLearning education platform. Most caregivers would have taken this module during competencies or orientation, but at various times. It will be taken by all participants in this study to serve as a baseline understanding of identifying and caring for patients at risk for falls. Participants will be enrolled in the module by a member of the research team, and learner transcripts will available through MyLearning education to confirm completion.

SUMMARY:
Falls place a huge financial burden on healthcare delivery systems, as well as physical and emotional harm to patients and families. Nurses are responsible for identifying fall risks and educating patients about fall risks and prevention, but first must have a thorough understanding of fall risk hazards themselves. The purpose of the study is to determine if enhanced education for caregivers using Virtual Reality simulation increases self-reported use of environmental fall risk interventions, and perceived effectiveness of those interventions, for caregivers on a medical-surgical unit. A secondary purpose is to explore the relationship between perceived effectiveness, unit norms, availability of resources, and self-reported behavior related to the use environmental interventions.

The study will use a matched-pair, clustered randomized controlled trial design. The setting is eight medical-surgical units across four hospitals. Unit-pairs at each hospital will be randomly assigned to control or intervention group. The sample will consist of clinical registered nurses and patient care nursing assistants. All participants will receive standard online fall risk education. Participants from the intervention units will also complete virtual reality simulation education delivered via an app on an iPhone that is attached to a headset. The Injurious Fall Risk Factors and Fall Prevention Interventions Survey will be used at baseline, 1 month post-, and 3 months post-education to measure perceived effectiveness, self-reported use, unit peer use, and availability of resources for use of environmental fall prevention interventions. A sample size of 30 participants per nursing unit will be needed for 90% power to detect mean differences of at least 0.5 points between groups.

ELIGIBILITY:
Inclusion Criteria:

* part-time and full-time registered nurses (RNs), Assistant Nurse Managers (ANMs), and patient care nursing assistants (PCNAs);
* participants must have greater than 50% of work time in direct patient care

Exclusion Criteria:

* holds PRN (as needed) or float position
* newly employed or in orientation at the time of the study
* reported history of dizziness or motion sickness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline rating of self-reported use of environmental fall prevention interventions at 1 month and 3 months post intervention | baseline, 1 month after intervention, and 3 months after intervention
  Using the Injurious Fall Risk Factors and Fall Prevention Interventions Survey, Part II (Tzeng & Yin, 2013), caregivers are asked to rate 23 interventions for reducing falls or injuries using a 5-point likert scale. Self-reported use of environmental fall prevention interventions is measured by rating the frequency of each intervention used by the participant in his or her practice over the last 30 days (1=rarely, 2=occasionally, 3=sometimes, 4=often, 5=always, or NA=not applicable/no knowledge).

SECONDARY OUTCOMES:
Change from baseline rating of perceived effectiveness of environmental fall prevention interventions at 1 month and 3 months post intervention | baseline, 1 month after intervention, and 3 months after intervention
  Using the Injurious Fall Risk Factors and Fall Prevention Interventions Survey, Part II (Tzeng & Yin, 2013), caregivers are asked to rate 23 interventions for reducing falls or injuries using a 5-point likert scale. Perceived effectiveness of environmental fall prevention interventions is measured by rating the effectiveness of each of the 23 interventions for reducing falls or injuries (1=Never effective, 2=Occasionally effective, 3=Sometimes effective, 4=Often effective, 5=Always effective or NA=not applicable/no knowledge).

OTHER OUTCOMES:
Change from baseline rating of perceived unit norms for use of environmental fall prevention interventions at 1 month and 3 months post intervention | baseline, 1 month after intervention, and 3 months after intervention
  Unit norms for use of environmental fall prevention interventions is measured by rating the frequency that participants observe the use of each intervention by peers on the unit (1=rarely, 2=occasionally, 3=sometimes, 4=often, 5=always, or NA=not applicable/no knowledge).
Change from baseline rating of availability of resources to implement environmental fall prevention interventions at 1 month and 3 months post intervention | baseline, 1 month after intervention, and 3 months after intervention
  Availability of resources to implement environmental fall prevention interventions is measured by rating how often resources limit the implementation each intervention. (1=Never, 2=Occasionally, 3=Sometimes, 4=Often, 5=Always or NA=not applicable/no knowledge). Scores will be reversed coded for analysis.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cleveland Clinic Avon Hospital, Avon, Ohio
  - Cleveland Clinic Hillcrest Hospital, Mayfield Heights, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouldin EL, Andresen EM, Dunton NE, Simon M, Waters TM, Liu M, Daniels MJ, Mion LC, Shorr RI. Falls among adult patients hospitalized in the United States: prevalence and trends. J Patient Saf. 2013 Mar;9(1):13-7. doi: 10.1097/PTS.0b013e3182699b64. PMID 23143749
- [Background] Fehlberg EA, Lucero RJ, Weaver MT, McDaniel AM, Chandler AM, Richey PA, Mion LC, Shorr RI. Impact of the CMS No-Pay Policy on Hospital-Acquired Fall Prevention Related Practice Patterns. Innov Aging. 2017 Nov;1(3):igx036. doi: 10.1093/geroni/igx036. Epub 2018 Feb 2. PMID 29911187
- [Background] Florence CS, Bergen G, Atherly A, Burns E, Stevens J, Drake C. Medical Costs of Fatal and Nonfatal Falls in Older Adults. J Am Geriatr Soc. 2018 Apr;66(4):693-698. doi: 10.1111/jgs.15304. Epub 2018 Mar 7. PMID 29512120
- [Background] Clyburn TA, Heydemann JA. Fall prevention in the elderly: analysis and comprehensive review of methods used in the hospital and in the home. J Am Acad Orthop Surg. 2011 Jul;19(7):402-9. doi: 10.5435/00124635-201107000-00003. PMID 21724919
- [Background] Haerling KA. Cost-Utility Analysis of Virtual and Mannequin-Based Simulation. Simul Healthc. 2018 Feb;13(1):33-40. doi: 10.1097/SIH.0000000000000280. PMID 29373382
- [Background] Hemming K, Girling AJ, Sitch AJ, Marsh J, Lilford RJ. Sample size calculations for cluster randomised controlled trials with a fixed number of clusters. BMC Med Res Methodol. 2011 Jun 30;11:102. doi: 10.1186/1471-2288-11-102. PMID 21718530
- [Background] Pottle J. Virtual reality and the transformation of medical education. Future Healthc J. 2019 Oct;6(3):181-185. doi: 10.7861/fhj.2019-0036. PMID 31660522
- [Background] Slade SC, Carey DL, Hill AM, Morris ME. Effects of falls prevention interventions on falls outcomes for hospitalised adults: protocol for a systematic review with meta-analysis. BMJ Open. 2017 Nov 12;7(11):e017864. doi: 10.1136/bmjopen-2017-017864. PMID 29133324
- [Background] Soong C, Shojania KG. Education as a low-value improvement intervention: often necessary but rarely sufficient. BMJ Qual Saf. 2020 May;29(5):353-357. doi: 10.1136/bmjqs-2019-010411. Epub 2019 Dec 16. No abstract available. PMID 31843878
- [Background] Tzeng HM, Yin CY. Most frequently observed risk factors for adult inpatient injurious falls in hospitals. Clin Nurse Spec. 2013 Nov-Dec;27(6):314-22. doi: 10.1097/NUR.0b013e3182a87271. PMID 24107755
- [Background] Tzeng HM, Yin CY. Most and least helpful aspects of fall prevention education to prevent injurious falls: a qualitative study on nurses' perspectives. J Clin Nurs. 2014 Sep;23(17-18):2676-9. doi: 10.1111/jocn.12295. Epub 2013 Jul 2. No abstract available. PMID 23815367
- [Background] Wan X, Wang W, Liu J, Tong T. Estimating the sample mean and standard deviation from the sample size, median, range and/or interquartile range. BMC Med Res Methodol. 2014 Dec 19;14:135. doi: 10.1186/1471-2288-14-135. PMID 25524443